CLINICAL TRIAL: NCT04247503
Title: Cohort Study of Pancreatic Cancer Risk
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-010791; U01CA210138 (NIH); NCI-2023-05521 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-01-23; First posted 2020-01-30 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Familial Pancreatic Cancer
MeSH Terms: conditions — Pancreatic carcinoma, familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 50 cc of blood annually for 5 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed to develop a cohort of individuals without pancreatic cancer, but who are at increased risk of developing it due to family history or genetic predisposition. These high-risk individuals will be asked to provide baseline and annual (serial) follow-up blood samples for the duration of the study funding. Mayo Clinic is part of a national Pancreatic Cancer Detection Consortium (PCDC)[1] which aims to establish a high-risk cohort with the goal of validating blood biomarkers (discovered/developed outside of this protocol) using the samples collected serially (annually) that predict or detect pancreatic cancer prior to clinical diagnosis.

DETAILED DESCRIPTION:
The high mortality rate of pancreatic cancer is primarily due to the advanced stage at diagnosis in the majority of cases. The five-year survival rate for this cancer is only 9%, the poorest survival rate of any major cancer, making pancreatic cancer the third leading cancer killer that affects both men and women in the United States. Five-year survival can be improved if the cancer is detected earlier.[2] It is thus important to apply cancer genetics, risk assessment, and early detection that can identify a population of high-risk individuals who can benefit from early detection.

A key strategy for effective early detection research in pancreatic cancer is to identify and build longitudinal high-risk cohorts and maintain data from baseline to follow up, and biobanking of repeated (annual) non-invasive biospecimen collections. The research to be performed would compare samples of participants who develop cancer over time compared to those who do not. Tests that would be applied to the biospecimen collections would use subsets of participants in designs that would provide the maximum amount of information about the performance of the assays in predicting who has cancer at an early stage [3,4].

The collection of biosamples and data for the family-based biobank resource/registry proposed here is partially funded by NCI funded U01 grants, through the PCDC [1]. At Mayo Clinic, NCI grant U01 CA210138 is the funding source. The PCDC is committed to developing a longitudinal cohort (registry) of individuals and family members currently without pancreatic cancer, but who are at high risk due to family history of pancreatic cancer or predisposition gene mutation status. High-risk individuals will be recruited at each site, and biospecimens will be logged, stored, administered, and studied by consensus protocols of members of the PCDC. The maintenance of protocols will be maintained by the PCDC Administrative Core at Mayo Clinic. The PCDC cohort will require a long-term investment and will be most successful with multiple contributing sites.

ELIGIBILITY:
Inclusion Criteria:

1. An individual who has previously consented to the Biospecimen Resource for Pancreas Research (Substudy #2 Family Studies) - IRB 355-06
2. Individual who does not have a personal history of pancreatic cancer and meets one of the following:

   1. Has relatives in family that contains pancreatic cancer, and carries a known germline mutation in APC, ATM, BRCA1, BRCA2, CDKN2A, EPCAM, MLH1, MSH2, MSH6, PALB2, PMS2, STK11, or TP53.

      OR
   2. Is a first- or second-degree blood relative of an individual with a diagnosis of pancreatic ductal adenocarcinoma (PDAC) and this PDAC patient has a germline mutation in APC, ATM, BRCA1, BRCA2, CDKN2A, EPCAM, MLH1, MSH2, MSH6, PALB2, PMS2, STK11, or TP53.

      OR
   3. Is a first- or second-degree blood relative of an individual with a germline mutation in one of these genes and where the mutation carrier is also a first-degree relative to a PDAC case.

      OR
   4. Is a blood relative to a PDAC patient in a family that contains three blood relatives (all maternal side or all paternal side) with PDAC.
3. Age

   1. 50 or older, OR
   2. Or within 10 years of the age of diagnosis of the youngest PDAC blood relative.
4. Individual with a valid United States mailing address. -

Exclusion Criteria:

1. Individual who has a personal history of PDAC
2. Individual who has received a bone marrow transplant, who has had a blood transfusion within the last 7 days, or who has an active hematologic malignancy (i.e., leukemia or lymphoma).
3. Individual who is unable to sign the informed consent because of mental incompetency or psychiatric illness
4. Individual who is non-English speaking
5. Individual who is a prison inmate -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals aged 50 and older without pancreatic cancer who are members of kindreds containing three blood relatives with pancreatic cancer, OR who carry a mutation in a known predisposition gene for pancreatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of cancer in the risk cohort | Through study completion, an average of 5 years.
  Enumeration of number of new cases of pancreatic cancer and other cancers that incidentally develop from baseline enrollment among those who enroll in the cohort. This number will be a numerator for a risk ratio. The denominator will be person years at risk starting from age 50.

SECONDARY OUTCOMES:
Association of baseline patient characteristics with incident cancers | through study completion an average of 5 years.
  Participants will complete questionnaires seeking demographic, clinical and family history, and exposures at baseline. We will evaluate by association studies (comparing participants with incident cancer to those who do not develop cancer) in order to discover various characteristics that may be associated with development of cancer. Specific characteristics that will be assessed (comparing participants who develop cancer to those who do not) include age at diagnosis of prevalent cancers, sex, personal history of diabetes, and family history (first and second degree) of pancreatic cancer and other cancers.
Measurement of test accuracy of biomarkers to detect pancreatic cancer | Through study completion, an average of 5 years.
  Biospecimens collected from patients will be used to assess the performance of potential biomarkers in detecting early pancreatic cancer. Two biomarkers that will be evaluated include serum CA19-9, fasting blood glucose and/or hemoglobin A1C. Additional biomarkers will be proposed and approved by scientific review in the future. We will compare samples collected longitudinally (prior to cancer diagnosis) from participants who develop cancer, to participants who do not develop cancer, and estimate test sensitivity and performance.

CONTACTS AND LOCATIONS:
Overall Officials: Shounak Majumder, M.D., Principal Investigator — The Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT04247503/ICF_000.pdf